CLINICAL TRIAL: NCT02150707
Title: The Differential Effects of Diabetes Therapy on Inflammation
Status: Completed | Type: Observational
Sponsor: University College Dublin (Other)
Collaborators: Irish Endocrine Society (Other); Royal College of Physicians (Other); Merck Sharp & Dohme LLC (Industry); Eli Lilly and Company (Industry)
Responsible Party: Principal Investigator, Karl Neff, Clinical Research Fellow, University College Dublin
Other Study IDs: DPP4201401
Record Dates: First submitted 2014-05-27; First posted 2014-05-30 (Estimated); Last update posted 2016-05-18 (Estimated); Status verified 2016-05

CONDITIONS: Diabetic Nephropathy; Type 2 Diabetes
MeSH Terms: conditions — Diabetic Nephropathies; Diabetes Mellitus, Type 2 | interventions — Dipeptidyl-Peptidase IV Inhibitors; Glucagon-Like Peptide 1; Liraglutide; Exenatide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Dipeptidyl-Peptidase IV Inhibitors: Newly started on DPP4 inhibitor for hyperglycaemia
  Interventions: Drug: Dipeptidyl-Peptidase IV Inhibitors
- Glucagon-Like Peptide 1: Newly started on GLP-1 for hyperglycaemia or obesity
  Interventions: Drug: Glucagon-Like Peptide 1

INTERVENTIONS:
Drug: Dipeptidyl-Peptidase IV Inhibitors — Dipeptidyl-Peptidase IV Inhibitors to treat hyperglycaemia
  Other Names: DPP4 inhibitors
  Groups: Dipeptidyl-Peptidase IV Inhibitors
Drug: Glucagon-Like Peptide 1 — Glucagon-Like Peptide 1 to treat hyperglycaemia
  Other Names: Liraglutide; Exenatide
  Groups: Glucagon-Like Peptide 1

SUMMARY:
This study aims to determine if different diabetes treatments have different effects on inflammation; in particular, kidney inflammation. This type of inflammation is common in people with diabetes, and can lead to kidney failure. This study will investigate the effect of different types of diabetes treatment on kidney inflammation. This will help us to decide if certain types of medicine should be preferred in people with evidence of inflammation in their kidneys, as this may help prevent major complications including kidney failure.

DETAILED DESCRIPTION:
In this prospective cohort study, patients who are clinically determined to require escalation of their glycaemic therapy, and prescribed a DPP4 inhibitor, GLP-1 receptor agonist, or insulin, will be invited to participate.

Blood and urine samples will be taken before, 4 to 8 weeks after, and 26 weeks after starting the new therapy. Markers of inflammation, renal function and glycemic control will be measured at each timepoint.

ELIGIBILITY:
Inclusion Criteria:

* Age over 30 years
* Diagnosis of type 2 diabetes for one year or more
* Diagnosis of DKD as defined by two distinct albumin:creatinine ratio measurements above the gender specific range in the local reference laboratory with an interval of no less than eight week between measurements
* Stable dose of an inhibitor of the renin angiotensin system for a period of 8 weeks

Exclusion Criteria:

* Any cognitive impediment that preclude the participant from giving free and informed consent
* Substance abuse including alcohol excess
* Use of a GLP-1 analogue in the last 6 months
* Pregnancy
* Hypersensitivity to the prescribed treatment

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will be a prospective cohort study with 120 participants: 40 per group. I have calculated this sample size to achieve a 90% power based on a 50% reduction in urinary chemokines and circulating pro-inflammatory immune cells 1-4. This power calculation anticipates a 10% dropout rate.
  Patients with DKD presenting to the diabetes service of St Vincent's University Hospital (SVUH) and Mater Misericordiae University Hospital (MMUH) who are commenced on GLP-1, DPP4i or insulin for the first time will be invited to participate in the study.
Sampling Method: Non-Probability Sample
Enrollment: 17 (Actual)
Dates: Start 2014-05; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Monocyte:chemoattractant protein 1 (MCP-1):creatinine ratio | 6 months

SECONDARY OUTCOMES:
Albumin:creatinine ratio | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Donal O'Shea, MD FRCPI, Study Director — University College Dublin; Carel W le Roux, PhD MB FRCP, Study Director — University College Dublin; Mensud Hatunic, MD MRCPI, Study Director — University College Dublin
Locations (1):
- Mater Misericordiae University Hospital, Dublin, Ireland

REFERENCES:
- [Background] Fenske WK, Dubb S, Bueter M, Seyfried F, Patel K, Tam FW, Frankel AH, le Roux CW. Effect of bariatric surgery-induced weight loss on renal and systemic inflammation and blood pressure: a 12-month prospective study. Surg Obes Relat Dis. 2013 Jul-Aug;9(4):559-68. doi: 10.1016/j.soard.2012.03.009. Epub 2012 Apr 10. PMID 22608055
- [Background] Hogan AE, Gaoatswe G, Lynch L, Corrigan MA, Woods C, O'Connell J, O'Shea D. Glucagon-like peptide 1 analogue therapy directly modulates innate immune-mediated inflammation in individuals with type 2 diabetes mellitus. Diabetologia. 2014 Apr;57(4):781-4. doi: 10.1007/s00125-013-3145-0. Epub 2013 Dec 21. PMID 24362727
- [Background] Hattori S. Sitagliptin reduces albuminuria in patients with type 2 diabetes. Endocr J. 2011;58(1):69-73. doi: 10.1507/endocrj.k10e-382. Epub 2010 Dec 28. PMID 21206136
- [Background] Wu JD, Xu XH, Zhu J, Ding B, Du TX, Gao G, Mao XM, Ye L, Lee KO, Ma JH. Effect of exenatide on inflammatory and oxidative stress markers in patients with type 2 diabetes mellitus. Diabetes Technol Ther. 2011 Feb;13(2):143-8. doi: 10.1089/dia.2010.0048. PMID 21284481